CLINICAL TRIAL: NCT03902548
Title: A Positron Emission Tomography (PET) Study to Compare the [18F]P16-129 and [18F]Florbetapir for Investigations of Amyloid β Pathology in Subjects With Alzheimer's Disease and Investigate the Biokinetics, Radiation Dosimetry, and Safety of [18F]P16-129 in Healthy Volunteers
Brief Title: Initial Investigation of [18F]P16-129 in Alzheimer's Disease Patients and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Five Eleven Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: JH-147896
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — (18 F)D3FSP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brain uptake and kinetics in Alzheimer's patients (Experimental)
  Interventions: Drug: [18F]P16-129
- Dosimetry in healthy volunteers (Experimental)
  Interventions: Drug: [18F]P16-129

INTERVENTIONS:
Drug: [18F]P16-129 — Injection of < 10 mCi [18F]P16-129 followed by PET/CT scanning
  Other Names: [18F]D3FSP

SUMMARY:
This study investigates the initial safety profile of [18F]P16-129 in healthy volunteers including dosimetry determination, and compares the uptake and kinetics of [18F]P16-129 with the FDA approved drug [18F]florbetapir in the brains of Alzheimer's disease patients.

ELIGIBILITY:
Part I - Brain uptake in Alzheimer's patients

Inclusion Criteria

1. Signed and dated written informed consent. Capacity for consent will be determined using the Alzheimer's Association Guidelines, developed at Johns Hopkins and described in Alzheimer's Association

   Consensus Recommendation: Research consent for cognitively impaired adults:

   Guidelines for Institutional Review Boards and Investigators (Alzheimer's Association 2004).
2. Have a study partner able to accompany the subject to all visits and answer questions about the subject.
3. Male or female, > 50 years of age
4. Have a diagnosis of probable AD, according to the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association criteria
5. The patient has a Mini Mental State Examination (MMSE) score at screening of at least 15 and no greater than 26.
6. Female patients must have had her last natural menstruation at least ≥24 months prior to the Screening Visit or have been surgically sterilized prior to the Screening Visit. Male patients must use two methods of contraception in combination if his female partner is of childbearing potential; OR have been surgically sterilized prior to the Screening Visit.
7. In the opinion of the investigator based on medical history and physical examination, can safely tolerate tracer administration and the scanning procedures.

Exclusion Criteria:

1. History or presence of a significant neurological diagnosis (other than AD) that may influence the outcome or analysis of the scan results; examples include but are not limited to stroke, traumatic brain injury, space occupying lesions, major head trauma, and Parkinson's disease.
2. History or presence of any clinically relevant hematological, hepatic, respiratory, cardiovascular, renal, metabolic, endocrine, or CNS disease or other medical conditions that are not well controlled, may put the subject at risk, could interfere with the objectives of the study, or make the subject unsuitable for participation in the study for any other reason in the opinion of the principal investigator.
3. The patient has a history of seizures, with the exception of childhood febrile seizures.
4. History of positive HIV, hepatitis B surface antigen (HBsAg), or hepatitis C virus / antibodies (anti-HCV)
5. Clinically relevant pathological findings in physical examination, ECG, vital signs, or laboratory values at the screening assessment that could interfere with the objectives of the study.
6. Have current clinically significant cardiovascular disease. The patient has, at the Screening Visit: an abnormal ECG that is, in the investigator's opinion, clinically significant, a QTcF > 470 ms.
7. Has had or is planning to have exposure to ionizing radiation that in combination with the study-related tracer administrations and scanning procedures would result in a cumulative exposure that exceeds recommended exposure limits.
8. Contraindications of MRI. Incidental findings on MRI scans that are pathognomonic for an active disease or pathological process which requires medical intervention will be exclusionary.
9. History of, or suffers from, claustrophobia or feels that he or she will be unable to lie still on their back in the MRI or PET scanner.
10. Patients who have received an investigational medication within the last 30 days. Additionally, the time between the last dose of the previous experimental medication and enrollment (completion of screening assessments) must be at least equal to 5 times the terminal half-life of the previous experimental medication.

Part II - Dosimetry in Healthy Volunteers

Inclusion Criteria

1. Healthy non-smoking males and females, as determined by medical history, physical examination, vital signs, clinical laboratory tests, and an electrocardiogram.

   1.1 Male subjects and their child bearing potential partners must be willing to use a reliable method of birth control for the duration of the study.

   1.2 Female subjects who are of childbearing potential must agree to use an adequate method of contraception for the duration of the study.
2. Between 18-45 years old, inclusive.
3. BMI between 18-30 kg/m2 inclusive.
4. Have clinical laboratory test results within the reference ranges for the population or results within acceptable deviations that are not considered by the investigator to be clinically significant.
5. All subjects and their partners of childbearing potential must commit to use two methods of contraception, one of which must be a barrier method, from the time of screening and throughout the study and until follow-up.
6. Less than 195 cm (6 feet and 5 inches) tall in order to accommodate the whole body scanning.
7. Have sufficient venous access.

Exclusion Criteria:

1. Are currently enrolled in or discontinued within the last 30 days from a clinical trial involving an investigational drug or device (other than the study drug) or are currently enrolled in any other type of medical research.
2. Are currently experiencing neuropsychiatric illness or severe systemic disease based on history and physical exam.
3. Have participated in other research protocols in the last year such that radiation exposure would exceed the annual limits.
4. Pregnant or nursing women.
5. History of head trauma with prolonged loss of consciousness (>10 minutes) or any neurological condition including stroke or seizure (excluding childhood febrile seizure) or history of migraine headache.
6. History of any clinically relevant hematological, hepatic, respiratory, cardiovascular, renal or CNS disease or other medical condition that is capable of constituting a risk factor when taking the study drug.
7. Suffer from claustrophobia and would be unable to undergo PET scanning.
8. Any confirmed significant allergic reactions against any drug, or multiple allergies.
9. Currently uses prescription medications, over-the-counter drugs or herbal remedies such as St. Johns Wort) which cannot be discontinued 14 days (or < 5 half-lives, whichever is longer), prior to the PET scan and throughout the study. Exceptions include daily multiple vitamins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-11-02 (Actual); Study Completion 2019-11-02 (Actual)

PRIMARY OUTCOMES:
Regional brain uptake of [18F]P16-129 and [18F]florbetapir | 30 - 90 minutes post injection
  Quantitative estimates of amyloid distribution in brain - SUV and SUVR
Cumulative organ [18F]P16-129 activity for estimates of radiation absorbed dose and effective dose | 0 - 240 min post injection
  dosimetry

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Alexoff D, Wong DF, Kuwabara H, Dannals RF, Ploessl K, Kung HF. Head to head comparison of two PET/CT imaging agents, [18F]D3FSP ([18F]P16-129) and [18F]AV45, in patients with alzheimer's disease. EJNMMI Res. 2025 Jun 22;15(1):77. doi: 10.1186/s13550-025-01276-w. PMID 40544409